CLINICAL TRIAL: NCT02397759
Title: Analysis of Cerebral Spinal Fluid and Plasma After Aneurysmal Subarachnoid Hemorrhage by Evaluating a Metabolomic Profile and the Proteasic Activity as Biomarkers for Early Detection of Arterial Vasospasm
Brief Title: Metabolomic Profile and Proteasic Activity as Biomarkers for Early Detection of Arterial Vasospas in Arterial Vasospasm After Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-54; 2013-A00184-41 (Registry Identifier: Ansm)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Subarachnoid Hemorrhage (SAH) From Ruptured Aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with severe SAH and vasospasm (Experimental): Patients with severe SAH from ruptured aneurysm requiring the establishment of an external ventricular derivation (EVD) and presenting vasospasm
  Interventions: Other: Blood draw and cerebrospinal fluid draw
- Patients with severe SAH without vasospasm (Experimental): Patients with severe SAH from ruptured aneurysm requiring the establishment of an external ventricular derivation (EVD) without vasospasm
  Interventions: Other: Blood draw and cerebrospinal fluid draw
- Patients with severe SAH without external ventricular derivati (Active Comparator): Patients with severe severe SAH from ruptured aneurysm without necessitating a EVD subarachnoid hemorrhage
  Interventions: Other: Blood draw and cerebrospinal fluid draw

INTERVENTIONS:
Other: Blood draw and cerebrospinal fluid draw

SUMMARY:
The subarachnoid hemorrhage (SAH) from ruptured aneurysm is a situation that is life-threatening, which is largely dependent on the occurrence of vasospasm from the 4th day after the bleeding. This vasopasm is responsible of clinical morbidity in 30 to 50% of patients. It occurs in 40% of patients with severe SAH.

Despite knowing this, the clinician has no biomarker for identifying patients at risk.

The project presented is original and includes a screening method without a priori to identify predictive biomarkers of vasospasm, likely to become therapeutic targets. In secondary objective we will focus on the protease activity of cerebrospinal fluid (CSF) and blood as a biomarker potential of vasoconstriction at the waning of subarachnoid hemorrhage.

This study will take place over a year prospectively. The inclusion of patients will be in the SAR 1 Hospital of Timone. Patients with severe severe SAH by rupture requiring the establishment of an external ventricular derivation (EVD) will be divided into two groups and compared to one group of patients without necessitating a EVD subarachnoid hemorrhage.

* Group 1: Patients with vasopasm
* Group 2: Patient presenting no vasopasm Detection of vasopasm was defined using a consensual definition. CSF samples (through EVD) and blood will be made upon arrival of the patient in intensive care and then between the 3rd and 4th day.

As the main criterion, we will identify biomarkers of vasospasm in blood and CSF without a priori assumption by metabolomics. Analysis will be by chromatography system coupled to a high resolution mass spectrometer. This method does not justify effective calculation because it is a step of generating hypotheses requiring further biological validation based on the identified targets.

The secondary criteria, we will study in the blood and CSF association between matrix metalloproteinases (MMP) 2 and 9 and the occurrence of vasopasm.

RESULTS: After comparative analysis of groups 1 and 2 in two phases of the study, we will define a metabolic profile that could identify predictive biomarkers vasopasm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe severe SAH by rupture requiring the establishment of an external ventricular derivation (EVD) will be divided into two groups
* Group 1: Patients with vasopasm
* Group 2: Patient presenting no vasopasm

Exclusion Criteria:

* Patients presenting an infectious or carcinologic meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
biomarkers iendtification of vasospasm | 3 years
  It will be identify biomarkers of vasospasm in blood and CSF without a priori assumption by metabolomics. Analysis will be by chromatography system coupled to a high resolution mass spectrometer

SECONDARY OUTCOMES:
occurrence of vasopasm | 3 years
  It will be study in the blood and CSF association between matrix metalloproteinases (MMP) 2 and 9 and the occurrence of vasopasm

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Hôpiital de la TIMONE ASSISTANCE PUBLIQUE HOPITAUX de MARSEILLE, Marseille, France

REFERENCES:
- [Derived] Chikh K, Tonon D, Triglia T, Lagier D, Buisson A, Alessi MC, Defoort C, Benatia S, Velly LJ, Bruder N, Martin JC. Early Metabolic Disruption and Predictive Biomarkers of Delayed-Cerebral Ischemia in Aneurysmal Subarachnoid Hemorrhage. J Proteome Res. 2024 Jan 5;23(1):316-328. doi: 10.1021/acs.jproteome.3c00575. Epub 2023 Dec 26. PMID 38148664
- [Derived] Triglia T, Mezzapesa A, Martin JC, Verdier M, Lagier D, Dufour H, Bruder N, Alessi MC, Velly LJ. Early matrix metalloproteinase-9 concentration in the first 48 h after aneurysmal subarachnoid haemorrhage predicts delayed cerebral ischaemia: An observational study. Eur J Anaesthesiol. 2016 Sep;33(9):662-9. doi: 10.1097/EJA.0000000000000494. PMID 27355865